CLINICAL TRIAL: NCT05278442
Title: Retrospective Evaluation of the Accuracy and Safety of the LaserArcs Femtosecond Cataract Surgery Arcuate Incision Nomogram in Patients Undergoing Cataract Surgery and Astigmatism Reduction
Brief Title: Evaluation of the Accuracy & Safety of the LaserArcs Nomogram
Status: Completed | Type: Observational
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2109 LaserArc
Record Dates: First submitted 2022-02-03; First posted 2022-03-14 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: LaserArc — LaserArcs.com is an online arcuate incision nomogram calculator initially developed on the basis of 12 months of data tabulation of patients undergoing femtosecond surgery with arcuate incisions

SUMMARY:
Evaluation of the Accuracy and Safety of the LaserArcs Femtosecond Cataract Surgery Arcuate Incision Nomogram in Patients Undergoing Cataract Surgery and Astigmatism Reduction

DETAILED DESCRIPTION:
Femtosecond lasers allow the precise placement of arcuate keratotomy incisions in patients undergoing cataract surgery. Though these surgical devices have been available for several years, most current nomograms designed to reduce astigmatism with these incisions are derived from those developed for metal or diamond knives. Anecdotal reports from surgeons indicate that the previous nomograms have limited accuracy in the setting of femtosecond laser surgery.

LaserArcs.com is an online arcuate incision nomogram calculator initially developed on the basis of 12 months of data tabulation of patients undergoing femtosecond surgery with arcuate incisions. since that time, its user base has grown because of the high accuracy its model provides. Currently over 3500 calculations are performed each month on this platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cataract and otherwise healthy eyes, not exhibiting any significant ocular morbidity that would be expected to influence outcome measures.
* Patients who are 22 years of age or older
* Patients whose preoperative astigmatism was greater than 0.5 D
* Patients who were implanted with a non-toric IOL.
* Patients whose laser astigmatic keratotomy was planned using the LASER arcs nomogram

Exclusion Criteria:

* Patients with visually significant co-morbidities (corneal, retina, optic nerve disease) that could affect their satisfaction with surgery
* Patients with surgical complications either during or after surgery (capsule tears, iris trauma, decentered IOL, cystoid macular edema, etc.) that would, in the judgment of the investigator, influence the outcome measures of the study.
* Patients with previous refractive surgery within the past 6 months prior to cataract surgery

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study aims to enroll 50 patients that had previous cataract surgery performed with femtosecond lasers.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint -Postoperative magnitude of manifest astigmatism (diopters) divided by preoperative magnitude of manifest astigmatism (diopters) | Up to 3 months
  Percent change in absolute magnitude of astigmatism

SECONDARY OUTCOMES:
Mean Attempted vs Achieved Correction (see description) | Up to 3 months
  Mean attempted vs achieved correction. Attempted correction=postop target astigmatism-pre-op corneal astigmatism), achieved correction=postop manifest cylinder-pre-op corneal astigmatism, attempted vs achieved=achieved correction-attempted correction mean attempted vs achieved=average of all individual calculated values for attempted vs achieved correction
Secondary Endpoint - Standard deviation of attempted vs achieved correction = standard deviation of of all individual calculated values for attempted vs achieved correction | Up to 3 months
  Standard deviation of attempted vs number of achieved correction of corneal astigmatism.

OTHER OUTCOMES:
Exploratory Endpoint - Postoperative manifest refraction cylinder and axis is the measured magnitude of spherical and cylindrical refraction at the postoperative visit. | Up to 3 months
  Postoperative manifest refraction for sphere, cylinder, and axis.

CONTACTS AND LOCATIONS:
Locations (1):
- Quantum Vision Centers, Belleville, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided